CLINICAL TRIAL: NCT03267407
Title: Vietnam Cryptococcal Retention in Care Study (CRICS) - Version 2.1
Brief Title: Vietnam Cryptococcal Retention in Care Study - Version 2.1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Principal Investigator, Vu Quoc Dat, Lead Coordinator, National Hospital for Tropical Diseases, Hanoi, Vietnam
Other Study IDs: 5U01GH000758-03 (NIH)
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: HIV/AIDS; Cryptococcal Meningitis; Opportunistic Infections, HIV Related; Cryptococcosis; Mycosis; Opportunistic; Mycosis Fungoides
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningitis, Cryptococcal; AIDS-Related Opportunistic Infections; Cryptococcosis; Mycoses; Mycosis Fungoides | interventions — Fluconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CrAg(+) and CM(-): (1) Patients with CrAg positive without meningitis results will receive preemptive high-dose fluconazole to prevent developing meningitis.
  Interventions: Other: Preemptive high-dose Fluconazole
- CrAg(+) and CM(+): (2) Patients with CrAg positive and meningitis results will receive standard treatment for cryptococcal meningitis, following national guidelines.
  Interventions: Other: Preemptive high-dose Fluconazole
- CrAg(-): (3) Patients with CrAg negative results will be managed as other HIV infected patients with the standard of care, following national guidelines.
  Interventions: Other: Preemptive high-dose Fluconazole

INTERVENTIONS:
Other: Preemptive high-dose Fluconazole — Patients with advanced HIV diseases are screened for Cryptococcal Antigen using LFA CrAg tests. Then patients with CrAg positivity and without meningitis are given preemptive high-dose fluconazole to prevent the development of cryptococcal meningitis, which is one of the leading cause of death among immunocompromized patients.
  Other Names: Preemptive Fluconazole

SUMMARY:
This is a multicenter prospective cohort evaluation of the implementation of a cryptococcal antigen (CrAg) screening program at selected outpatient HIV clinics (OPCs) and network laboratories in Vietnam.

DETAILED DESCRIPTION:
The project will be implemented in 2 phases; Phase 1: From August 2015 to March 2017 [projected], HIV-infected patients who present for HIV care and undergo CD4 testing will be reviewed to determine the proportion of newly presenting patients with advanced disease (CD4 ≤100 cells/μL). Reflex CrAg screening will be performed using Lateral Flow Assay (LFA) for those with CD4≤100 cells/μL, per Vietnam national guidelines.

Patients with CD4≤100 cells/μL who present for antiretroviral treatment (ART) at a study OPCs-CRICS Sites- will be recruited into the longitudinal study and followed up with assessments and the collection of routine and supplemental data for 12 months or through September 2017 (whichever comes sooner). Those who are CrAg-positive, but have no features of central nervous system (CNS) disease, will be treated with high-dose fluconazole. Those with symptoms of CNS disease will be treated according to national guidelines. Survival, retention in care, and other clinical outcomes will be documented for patients who test CrAg-positive and are treated with fluconazole and those who test CrAg-negative. Data from those tested at participating labs but not eligible for enrollment in the longitudinal study will contribute to the estimation of the prevalence of CrAg.

Phase 2: From April 2017 to September 2017, a cost and cost-effectiveness analysis of CrAg screening will be conducted, a routine screening will be continued at existing sites and expanded to additional sites (preferentially to hospitals affiliated with Phase 1 OPCs and to other OPCs whose CD4 testing is conducted at laboratories already conducting CrAg screening as part of Phase 1). CrAg tests will also be made available to screen all patients with CD4≤100 cells/μL including those who are treatment-experienced. The test will also be made available for use among symptomatic patients for diagnostic purposes, including cerebral spinal fluid (CSF) and blood testing. Investigators will monitor prevalence at each testing site, but screened patients will not be enrolled in longitudinal follow-up. Phase 2 will last for at least 6 months based on the availability of funding and fluconazole for those who screen CrAg positive and the availability/stability of CD4 testing.

[Note that follow up of patients enrolled in Phase 1 will continue during this time period, but is considered to be part of Phase 1 rather than Phase 2. Also, sites included in Phase 2 may change over time as a result of the instability of CD4 testing (e.g., if participating laboratories stop conducting CD4 testing, those sites might no longer be included; if participating laboratories begin CD4 testing for other sites, those sites might be included).]

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years (having passed 18th birthday using Western calendar)
* Confirmed HIV infection using National Testing Algorithm
* CD4 ≤100 cells/μL
* Able to provide written informed consent
* Enrolled at and plan to receive ongoing outpatient care at one of the selected study OPCs

Exclusion Criteria:

* History of prior CM
* Receipt of systemic antifungal medication for more than 4 consecutive weeks within the past 6 months
* Receipt of ART for more than 4 consecutive weeks within the past year
* For CrAg-positive patients only: Known to be currently pregnant or planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HIV infection (CD4<100 cells/microliters) who are eligible to inclusion and exclusion criteria are recruited and followed up into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV-infected adults who have CD4 count ≤ 100 cells/μL | August 2015 to March 2017
  The number of HIV-infected adults with CD4 count ≤ 100 cells/μL divided by the total number of HIV-infected patients.
Prevalence of CrAg-positivity among HIV-infected patients with CD4 ≤100 cells/μL | August 2015 to March 2017
  The number of CrAg-positivity divided by the number HIV-infected patients with CD4 ≤100 cells/μL
Clinical outcomes including common causes of mortality for people living with HIV (PLHIV) with CD4 ≤ 100 cells/μL who are enrolled in a programmatic rollout of screening for CrAg | August 2015 to March 2017
  Clinical outcomes include HIV-related hospitalization, causes of death, new AIDS defining opportunistic infections at 6 and 12 month.
Twelve (12) month all-causes and cryptococcal meningitis (CM)-related mortality among patients who screen CrAg-positive and CrAg-negative | August 2015 to March 2017
  The 12-month mortality among two groups of HIV-infected patients with CD4 ≤ 100 cells/μL who are enrolled in care and treatment:
  * Those who are CrAg-positive and are treated with high-dose fluconazole;
  * Those who are CrAg-negative.

SECONDARY OUTCOMES:
Twelve (12) month retention among patients who screen CrAg-positive and CrAg-negative | August 2015 to March 2017
  The 12-month retention in care among two groups of HIV-infected patients with CD4 ≤ 100 cells/μL who are newly enrolled in care and treatment.
Challenges associated with implementation of routine plasma CrAg screening in clinics providing HIV care | August 2015 to March 2018
  The challenges associated with implementation may include lost to follow up, incomplete documentation, and poor retention in care.
Lessons learned with participating sites | August 2015 to March 2018
  This will be delivered at reflection and transition workshops with participating sites.
Total costs and unit cost per person screened, per CrAg+ treated by site, lab facility type, and cost component. | August 2015 to March 2017
  The costs of implementing CrAg screening based on data to be collected at 22 participating clinics participating in Phase 1 and provider costs associated with CM treatment.
Incremental cost-effectiveness ratio (cost per CM death averted and cost per quality adjusted life year (QALY)) | August 2015 to March 2017
  The incremental cost-effectiveness analysis of CrAg screening compared with a standard of care (no CrAg screening, and treatment for symptomatic CM only).
Total cost savings and amount of financial resources required to implement CrAg screening | August 2015 to March 2017
  Potential cost savings from implementing CrAg screening and financial resources required to implement CrAg screening under different scale-up scenarios and for national rollout
Proportion of stored samples that test positive for TmAg | August 2015 to March 2017
  The prevalence of Talaromyces marneffei antigenemia (TmAg) in stored CRICS samples using the Mannose phosphate isomerase 1 (MP1) enzyme-linked immunosorbent assay (ELISA)
Six (6) and twelve (12) month all-causes and Talaromyces marneffei-related mortality among patients who screen TmAg-positive and TmAg-negative | August 2015 to March 2017
  The impact of TmAg positivity on mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kinh V Nguyen, MD, Principal Investigator — National Hospital for Tropical Diseases, Hanoi, Vietnam
Locations (1):
- National Hospital for Tropical Diseases, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Please contact principal investigators for any inquiries.

DOCUMENTS (2):
  • Study Protocol (2017-01-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03267407/Prot_000.pdf
  • Informed Consent Form (2017-01-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03267407/ICF_001.pdf